CLINICAL TRIAL: NCT01625650
Title: The Corrona Effectiveness Registry to Study Therapies for Arthritis and Inflammatory Conditions Sub-study: The Corrona CERTAIN Sub-study
Brief Title: Effectiveness Registry to Study Therapies for Arthritis and Inflammatory Conditions: The Corrona CERTAIN Sub-study
Acronym: CERTAIN
Status: Completed | Type: Observational
Sponsor: CorEvitas (Network)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: New England IRB 02-021; NEIRB 02-021 (Registry Identifier: Corrona, LLC)
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2016-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Registry; RA; Biologic; Medications; Rheumatology
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood tests: at each study blood is obtained to examine, lipid levels with direct ( non fasting) LDL, a high sensitivity CRP as well as toxicity monitoring labs including a complete blood count and a comprehensive panel. During the baseline visit DNA is collected upon consent - to allow future genetic and pharmacogenetic studies- and also serology markers and immunoglobulin levels. During the first three visits RNA serum and plasma for storage and future experiments are collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rheumatology: Patients who present at enrolling sites across the US are invited to enroll if eligible.

SUMMARY:
The CORRONA CERTAIN Sub-study of the Consortium of Rheumatology Researchers of North America, Inc. is a Sub-study of the CORRONA Data Collection Program.

The CERTAIN Sub-study is designed to systematically collect and document use patterns, effectiveness, comparative effectiveness and safety of biologic agents used in the management of Rheumatoid Arthritis (RA).

DETAILED DESCRIPTION:
Biologic therapies (including biologic medications like Enbrel, Humira, Remicade, Cimzia, Simponi, Actemra, Rituxan and Orencia) have changed the treatment of RA, but the differences in safety and/or effectiveness of each biologic therapy are not all known. We are doing this study in order to try to see if one or more of these treatments are better than the others. The use of databases like the CORRONA Organization database gives us information that helps us to understand why such drugs are used, reasons for starting or stopping drugs, for whom they are prescribed, and to monitor changes in patients' abilities to perform daily activities and gather information on family or social history.

ELIGIBILITY:
Inclusion Criteria:

* The CORRONA CERTAIN Sub-study is particularly focused on understanding the effectiveness and safety of biologic medications. Male and female patients, who

  1. are at least 18 years of age;
  2. have a documented diagnosis of RA by their treating rheumatologist;
  3. have at least moderate disease activity; and
  4. are initiating a biologic agent that has not be used for their treatment in the past are eligible to participate.

     Moderate disease activity is defined by a CDAI score greater than 10.

     Exclusion Criteria:

     Disease other than RA that do not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ppproximately 3,000 subjects from 100 sites will participate in this Sub-study and that approximately 30, and up to 200, subjects from this site will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 2795 (Actual)
Dates: Start 2010-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Pappas, MD, MPH, Study Chair — CORRONA INC.
Locations (1):
- The Center For Rheumatoligy, Albany, New York, United States

REFERENCES:
- [Derived] Harrold LR, Bryson J, Lehman T, Zhuo J, Gao S, Han X, Schrader A, Rebello S, Pappas DA, Sommers T, Kremer JM. Association Between Baseline Anti-cyclic Citrullinated Peptide Antibodies and 6-Month Clinical Response Following Abatacept or TNF Inhibitor Treatment: A Real-World Analysis of Biologic-Experienced Patients with RA. Rheumatol Ther. 2021 Jun;8(2):937-953. doi: 10.1007/s40744-021-00310-2. Epub 2021 May 28. PMID 34047953
- [Derived] Harrold LR, Litman HJ, Connolly SE, Alemao E, Kelly S, Rebello S, Hua W, Kremer JM. Comparative Effectiveness of Abatacept Versus Tumor Necrosis Factor Inhibitors in Patients with Rheumatoid Arthritis Who Are Anti-CCP Positive in the United States Corrona Registry. Rheumatol Ther. 2019 Jun;6(2):217-230. doi: 10.1007/s40744-019-0149-3. Epub 2019 Mar 13. PMID 30868550
- [Derived] Pappas DA, John A, Curtis JR, Reed GW, Karki C, Magner R, Kremer JM, Shewade A, Greenberg JD. Dosing of Intravenous Tocilizumab in a Real-World Setting of Rheumatoid Arthritis: Analyses from the Corrona Registry. Rheumatol Ther. 2016 Jun;3(1):103-115. doi: 10.1007/s40744-016-0028-0. Epub 2016 Feb 8. PMID 27747515
- See also: CORRONA Inc. Web site — http://www.CORRONA.org